CLINICAL TRIAL: NCT03933579
Title: A Nation-wide Multicenter Registry and Biobank Program for Deep Phenotyping of Idiopathic and Hereditary Pulmonary Arterial Hypertension in Korea: the PAH Platform for Deep Phenotyping in Korean Subjects (PHOENIKS) Cohort
Brief Title: The PAH Platform for Deep Phenotyping in Korean Subjects
Acronym: PHOENIKS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Sejong General Hospital (Other); Chonnam National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Saint Vincent's Hospital, Korea (Other); Seoul National University (Other); Chungnam National University Hospital (Other); Wonju Severance Christian Hospital (Other); Asan Medical Center (Other); Wonkwang University Hospital (Other); Chungbuk National University Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); The Catholic University of Korea (Other); Seoul National University Bundang Hospital (Other); Pusan National University Hospital (Other); Chonbuk National University Hospital (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Wook-Jin Chung, Professor, Gachon University Gil Medical Center
Other Study IDs: WJC-IIT-1002
Record Dates: First submitted 2019-04-10; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Arterial Hypertension; Deep Phenotyping; Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Each participating hospitals will be collecting whole blood from each patient, through which DNA, RNA, serum, plasma, and peripheral blood mononuclear cells will be extracted from the buffy coat layer for further multi-omics analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Deep phenotyping — Each participating hospitals will be collecting whole blood from each patient, through which DNA, RNA, serum, plasma, and peripheral blood mononuclear cells will be extracted from the buffy coat layer for further multi-omics analysis.

SUMMARY:
A total of 16 regional hospitals will be registering clinical data and biological specimens of idiopathic pulmonary arterial hypertension (IPAH)/heritable pulmonary arterial hypertension (HPAH) patients across Korea. The diagnosis of pulmonary arterial hypertension(PAH) will be based on right heart catheterization, where PAH caused by etiology other than HPAH or IPAH will be excluded. All clinical data will be stored to a government-based online database. Each participating hospitals will be collecting whole blood from each patient, through which DNA, RNA, serum, plasma, and peripheral blood mononuclear cells will be extracted from the buffy coat layer for further multi-omics analysis.

DETAILED DESCRIPTION:
Study Objectives The current study is a multicenter registry and biobank based on South Korean populations to construct a database for the elucidation the molecular and genetic modifiers of PAH. The ultimate goal is to utilize deep phenotypic data for prognosis prediction and discovery of biomarkers and targeted therapies.

Study Sample The current study will initially exclude the most frequent form of PAH in Korea, the connective tissue disease (CTD)-related PAH, and focus on the diagnosis and deep phenotyping of idiopathic PAH (IPAH) and heritable PAH (HPAH) patients. The inclusion criteria are as follows: (1) over 18 years of age, (2) mean pulmonary arterial pressure of 25mmHg or higher confirmed by right heart catheterization (RHC), (3) pulmonary vascular resistance ≥ 240 dynes∙s∙cm-5, (4) left ventricle diastolic pressure (LVDEP) or pulmonary capillary wedge pressure (PCWP) ≤ 15mmHg. Exclusion criteria are: (1) patients with drug-induced-PAH, (2) CTD, human immunodeficiency virus (HIV) infection, portal hypertension, congenital heart disease, or Schistosomiasis associated-PAH, (3) long-term responders to calcium channel blockers, (4) PAH patients with overt features of venous capillaries involvement, leaving IPAH and HPAH patients among group 1 of PH to be evaluated. HPAH will be diagnosed by identifying patients with heterozygous pathogenic variants of predetermined genes such as BMPR2, ACVRL1, ENG, CAV1, SMAD1, SMAD4, SMAD9, KCNK3, and EIF2AK4. Patients without a specific genetic mutation will then be categorized as IPAH patients. The genomic data of family members across 3 pedigrees of an HPAH patient will also be analyzed. All clinical and biological data will be reported to a customized web-based case report form called the iCReaT system managed by the Korean Center for Disease Control. All collected biospecimens will be stored at the Korean National Institute of Health main storage. Although the current analysis is planned to be limited to IPAH and HPAH patients, our steering committee plans to expand to all types of PAH in subsequent studies. This study was approved by the institutional ethics committee of each participating institutions and complied with the Declaration of Helsinki (6th revision). An informed consent will be received by each patient.

Baseline Data and Biospecimen Collection The baseline data from the registered patients across the 16 regional hospitals will include the following: WHO functional classification, 6-minute walking test, blood sample, electrocardiogram, chest X-ray, echocardiography, optional pulmonary-cardio exercise test, optional Cardiac MRI, and RHC. Detailed information of each exams are specified in Table 2. The registered patient will be followed up on a regular basis for further data and biospecimen collection.

With the patient's blood sample, DNA, RNA, serum, plasma, and peripheral blood mononuclear cells (PBMC) from the buffy coat will be separated and be extracted for further storage and studies. For the DNA sample, 2.5ml of the whole blood will be stored in a PAX gene DNA tube at the collecting site, and it will be carried to the main center at 4~10 C. At the main center, it will, then, be transferred to a 2ml cryotube to be stored at -70~80C. For patient's RNA collection, 2.5 mL of whole blood will be collected at PAX gene RNA tube, and it will be sent to the main center at 4~10 C, which will also be further transferred to a cryotube to be stored at -70~80C.

Patient's serum, plasma and the buffy coat will also be collected. At the respective collection sites, serum will be collected at a serum separation tube, and after 30 minutes of venipuncture, it will be centrifuged and stored at -20C. For patient's plasma, cell preparation tube will be used within 2 hours of blood collection. Then, each sample will be ready to be stored at -20C by treating the samples with human serum type antibody, DMSO, and freezing medium. To separate and extract PBMC, white buffy coat layer will be separated and be stored at a 1.5ml tube with a freezing medium at -20C. The collected baseline data will then go through a clean-up process and further evaluation of its quality will be done. In addition, five patients will be selected to do a whole-genome sequencing. All the collected biospecimen will be donated to NIH center storage, and will be further used for a multi-omics studies in order to deep phenotype the patient's specimens.

Patient Follow Up All patients will be followed up twice or more a year, with expected 80% follow up rate. During the second and third year, patient registry and data collection will be continued with the same protocol. To maintain the credibility of collected data, the steering committee will continuously monitor and audit the collected data. Protocol may be further crafted after evaluating the previous year's data. In addition, effective data management strategies, including a guideline to standardize patient's body measurement and blood sample will be developed. Ten patient samples will be selected for a next generation sequencing, and we will be utilized in discovering novel genetic mutations.

Genetic Mutation Analysis across Three-Pedigrees for HPAH Patients In order to determine patients with HPAH, a familial genetic study will be performed. A three-generation pedigree for each PAH patient with with or without the existence of a BMPR2, ACVRL1, ENG, CAV1, SMAD1, SMAD4, SMAD9, KCNK3, and/or EIF2AK4 mutation will be evaluated. Blood samples from family members of patients with a HPAH will be collected for genetic screening.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Mean pulmonary arterial pressure of 25mmHg or higher confirmed by right heart catheterization (RHC)
* Pulmonary vascular resistance ≥ 240 dynes∙s∙cm-5
* Left ventricle diastolic pressure (LVDEP) or pulmonary capillary wedge pressure (PCWP) ≤ 15mmHg

Exclusion Criteria:

* Patients with drug-induced-PAH
* Patients with CTD, human immunodeficiency virus (HIV) infection, portal hypertension, congenital heart disease, or Schistosomiasis associated- PAH
* Long-term responders to calcium channel blockers
* PAH patients with overt features of venous capillaries involvement

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Idiopathic PAH and heritable PAH patients in Korea
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes of death and hospitalization | 3 years
  A composite of death and hospitalization

SECONDARY OUTCOMES:
6 minute walk test | 3 years
  6 minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Medicine, Gachon University, Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share data

REFERENCES:
- [Derived] Jang AY, Kim S, Park SJ, Choi H, Oh PC, Oh S, Kim KH, Kim KH, Byun K, Chung WJ; PHOENIKS Investigators. A Nationwide multicenter registry and biobank program for deep phenotyping of idiopathic and hereditary pulmonary arterial hypertension in Korea: the PAH platform for deep phenotyping in Korean subjects (PHOENIKS) cohort. Clin Hypertens. 2019 Sep 15;25:21. doi: 10.1186/s40885-019-0126-8. eCollection 2019. PMID 31534782